CLINICAL TRIAL: NCT02822521
Title: A Novel Mobile App & Population Management System to Manage Rheumatoid Arthritis Flares
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Daniel H. Solomon, M.D.,MPH, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014P002312
Record Dates: First submitted 2016-06-22; First posted 2016-07-04 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Arthritis; Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Mobile Health; Pain; Arthritis
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Application + Population Manager (Experimental): This arm of the study will contain half the study population after randomization. The participants in this arm will receive the mobile application with daily questions after the first visit. A population manager will review patient-reported symptoms via a web-base dashboard and contact the subject based on pre-specified guidelines.
  Interventions: Other: Mobile Application; Other: Population Management System
- No Mobile Application (No Intervention): This arm of the study will contain half the study population after randomization. The participants in this arm will not receive the mobile application after the first visit. Although participants will be provided with the contact information of a study staff member, there will be no active contact with the subject unless he/she initiates.

INTERVENTIONS:
Other: Mobile Application — A mobile health application that asks daily questions about participants' pain, function, and disease activity.
  Arms: Mobile Application + Population Manager
Other: Population Management System — Study staff will act as care managers behind a web-based dashboard to monitor participants' responses to the daily questions on the mobile application and connect them with their HCPs.
  Arms: Mobile Application + Population Manager

SUMMARY:
The overall objective of this proposal is to implement a smart phone application (app) + population management system to monitor rheumatoid arthritis (RA) disease activity between scheduled physician office visits. The population management system includes: 1) a web-based dashboard that consolidates incoming patient-reported data using pre-programmed algorithms to identify increases in disease activity, and 2) the population manager, a trained individual who monitors the web-based dashboard and connects patients with their healthcare providers (HCPs). The investigators central hypothesis is that the combined smart phone app + population management system will improve patient satisfaction and management of RA disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA by a board-certified rheumatologist
* Taking a DMARD (sulfasalazine, methotrexate, leflunomide, azathioprine, certolizumab, cyclosporine, adalimumab, etanercept, infliximab, golimumab, abatacept, tocilizumab, anakinra, tofacitinib, rituximab, hydroxychloroquine)
* Own a smart phone with either an Android or iPhone operating system
* Be English-speaking

Exclusion Criteria:

* Patients who do not plan on receiving follow-up care at the Brigham and Women's Hospital Arthritis Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2016-11; Primary Completion 2025-09 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire for Medication (TSQM) | 6 months
Clinical Disease Activity Index (CDAI) | 6 months
Perceived Efficacy in Patient-Physician Interactions Questionnaire (PEPPI) | 6 months

SECONDARY OUTCOMES:
Patient Activity Scale-II (PAS-II) | 6 months
Flare Assessment in Rheumatoid Arthritis (FLARE) questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YC, Lu F, Colls J, Luo D, Wang P, Dunlop DD, Muhammad LN, Song J, Michaud K, Solomon DH. Outcomes of a Mobile App to Monitor Patient-Reported Outcomes in Rheumatoid Arthritis: A Randomized Controlled Trial. Arthritis Rheumatol. 2021 Aug;73(8):1421-1429. doi: 10.1002/art.41686. Epub 2021 Jun 18. PMID 33559338
- [Derived] Colls J, Lee YC, Xu C, Corrigan C, Lu F, Marquez-Grap G, Murray M, Suh DH, Solomon DH. Patient adherence with a smartphone app for patient-reported outcomes in rheumatoid arthritis. Rheumatology (Oxford). 2021 Jan 5;60(1):108-112. doi: 10.1093/rheumatology/keaa202. PMID 32572490
- [Derived] Wang P, Luo D, Lu F, Elias JS, Landman AB, Michaud KD, Lee YC. A Novel Mobile App and Population Management System to Manage Rheumatoid Arthritis Flares: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 11;7(4):e84. doi: 10.2196/resprot.8771. PMID 29643053